CLINICAL TRIAL: NCT00350376
Title: Study on Asthma Treatments on Daily Activities as Reported by Patients (STAR)
Brief Title: Impact of Asthma Treatments on Daily Activities
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ovation Research Group (Industry)
Collaborators: Genentech, Inc. (Industry)
Other Study IDs: 1467
Record Dates: First submitted 2006-07-05; First posted 2006-07-10 (Estimated); Last update posted 2006-07-10 (Estimated); Status verified 2006-07

CONDITIONS: Asthma; Allergies
Keywords: asthma; allergies; Xolair; Advair
MeSH Terms: conditions — Asthma; Hypersensitivity

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Other

SUMMARY:
The primary objective of this web-based, cross-sectional study is to assess and compare the ability to sleep, work or go to school, and to participate in leisure activities among subjects who are receiving Xolair treatment and subjects who were eligible to receive Xolair, but instead have been using Advair for at least 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Have asthma and allergies
* Currently taking Xolair® or Advair®
* Started Xolair® treatment within the last 4 to 12 months OR have been taking Advair® for at least 12 months
* Between 18 and 55 years of age
* A non-smoker for at least 6 months
* Have internet access

Ages: 18 Years to 55 Years | Sex: All
Age Groups: Adult
Enrollment: 1500
Dates: Start 2006-06

CONTACTS AND LOCATIONS:
Overall Officials: Susan D Mathias, MPH, Principal Investigator — Ovation Research Group
Locations (1):
- Ovation Research Group, San Francisco, California, United States